CLINICAL TRIAL: NCT04219462
Title: Effect of Extracorporeal Shock Wave Therapy (ESWT) on Erectile Dysfunction in Type 2 Diabetes Mellitus Patients
Brief Title: Effect of ESWT on ED in Type 2 Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002577
Record Dates: First submitted 2020-01-01; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Erectile Dysfunction; Diabetes Mellitus, Type 2
Keywords: extracorporal shock wave
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 40 patients assigned to two groups
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): twenty men receive extracorporeal shock wave (ESWT) twice weekly for 3 consecutive weeks and repeated after a 3-week rest period, for a total of 12 treatment sessions. The patients will receive ESWT for 15 minutes at an energy level of 0.09 and a frequency of 120 shocks/min (1800 pulses per session). Shockwaves were delivered to the distal, mid, and proximal penile shaft, as well as to the left and right crura +sildenafil 5mg once daily for 3 months.
  Interventions: Device: active extracorporeal shock wave
- control group (Sham Comparator): twenty men will receive sham treatment underwent identical therapy with Extracorporal shock wave therapy (ESWT) application with a similar appearance and sound as the active low intensity extracorporal shock wave therapy (ESWT), although shock wave propagation to the tissue wills be blocked by a metal plate that will inserted into the sham applicator + sildenafil 5mg once daily for 3 months.
  Interventions: Device: sham extracorporeal shock wave

INTERVENTIONS:
Device: active extracorporeal shock wave — Ultrasound gel was used as a coupling agent, and the applicator of extracorpral shock wave therapy (ESWT) will be held perpendicular to the treatment surface throughout the treatment. Men in this group (n= 20) men receive ESWT twice weekly for 3 consecutive weeks and repeated after a 3-week rest period, for a total of 12 treatment sessions. The patients will receive ESWT for 15 minutes at an energy level of 0.09 and a frequency of 120 shocks/min (1800 pulses per session). Shockwaves were delivered to the distal, mid, and proximal penile shaft, as well as to the left and right crura + 5 mg sildnafil once daily for 3 months
  Arms: study group
Device: sham extracorporeal shock wave — twenty men will receive sham treatment underwent identical therapy with ESWT application with a similar appearance and sound as the active extracorporal shock wave therapy (ESWT), although shock wave propagation to the tissue wills be blocked by a metal plate that will inserted into the sham applicator + sildenafil 5mg once daily for 3 months.
  Arms: control group

SUMMARY:
Diabetes mellitus (DM) is known not only for its widespread prevalence, but also for its significant complications including cerebrovascular disease, coronary artery disease, renal failure, vision loss, and neuropathy. Of particular importance to sexual medicine, diabetes has also been strongly associated with erectile dysfunction (ED).ED is defined as the inability to obtain and/or maintain the erection firm enough to achieve a successful sexual intercourse on a regular basis. It is a more common condition in males with type 2 DM. In the field of sexual medicine numerous studies have shown that extracorporal shock wave therapy (ESWT) is safe, noninvasive, and, most importantly, an effective method for treating vascular ED

DETAILED DESCRIPTION:
ED in DM is often complex and caused by several mechanisms including vascular disease, autonomic neuropathy, hormonal imbalance, and psychogenic factors. However, as the endothelial dysfunction is an important factor contributing to the development of ED in diabetic patients, such patients can be resistant to phosphodiesterase 5 inhibitors (PDE5I) like sildenafil therapy. There are reports of lower efficacy of sildenafil in DM patients compared to general population.In the field of sexual medicine numerous studies have shown that ESWT is safe, noninvasive, and, most importantly, an effective method for treating vascular ED

Before starting the study, clearance will be obtained from the institutional ethical committee and prior informed consent of all the participants will be obtained before conducting the study. Patients will be recruited from outpatient clinic of andrology (Cairo University Hospitals). The patients were randomly divided into two equal groups:

Group (1): (Study group): Men in this group (n= 20) men receive extracorporeal shock wave (ESWT) twice weekly for 3 consecutive weeks and repeated after a 3-week rest period, for a total of 12 treatment sessions+sildenafil 5mg) Group (2): (Control group):) will receive sham treatment underwent identical therapy with ESWT application with a similar appearance and sound as the active low intensity ESWT+sildenafil 5mg

ELIGIBILITY:
Inclusion Criteria:

1. Forty married diabetic type 2 men with mild and moderate ED score (21-8) on Five-Item Version of the International Index of Erectile Function.
2. Patients who will have erectile dysfunction ( ED) from 6 months.
3. Patients with diabetes mellitus ( DM )duration ≥ 5 years with fasting blood glucose level of ≥ 126 mg/dl and glycosalyated haemoglobin (HbA1c ) ≥ 6.5% mg dl.
4. Body mass index ( BMI) will be < 30 kg/m²
5. The age of patients will be between 40- 60 years.

Exclusion Criteria:

* History of pelvic trauma, pelvic surgery, psychiatric disease.
* Patients with neuromuscular disorders, cardiovascular or pulmonary problems and spinal cord injuries.
* Vascular surgical intervention that recommended for the patients.
* Other renal conditions, respiratory disease, liver failure.
* Prostatectomy and patients with prostatic disease.
* Patients lacking complete follow-up data.
* hypogonadism.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
the Five-Version of International Index of Erectile function | 6 months after last treatment session
  Each patient will self- administrated the Arabic translated five- Item Version of International Index of Erectile Function (IIEF-5) (in which every patient in both groups will be asked about erectile dysfunction (ED) over their last four weeks). The procedure of IIEF-5 conducted in the following steps:
  1. The patient will be asked to answer each item by choosing an answer from the five answers of each five items
  2. The number opposite to each answer from the five answers will be determined
  3. The final number obtained by the sum of the ordinal responses to the five items.
  4. The improvement of erectile dysfunction will be detected according ED severity classification: no ED (score 25-22) mild ED (score 21-17), mild to moderate ED (score 16-12), moderate ED (score 11-8) and severe ED (score 7-1).
  5. Measurements will be done before initial session in both groups. Follow up will be after the sixth treatment and at 1, 3, 6 months in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Al shymaa s abdelazem, lecturer, Principal Investigator — lecturer of basic sciences- faculty of physical therapy- cairo university
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt